CLINICAL TRIAL: NCT06242977
Title: Efficacy of EMLA Cream Assisted Loco-sedation for Office-based Andrology Procedure: A Randomized Controlled Study
Brief Title: Efficacy of EMLA Cream Assisted Loco-sedation for Office-based Andrology Procedures
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Premal Patel, MD, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS25862 (H2023:047)
Record Dates: First submitted 2024-01-22; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Scrotum Disease; Hydrocele Male; Spermatocele; Scrotal Hematocele; Local Anesthesia
MeSH Terms: conditions — Spermatocele; Hematocele | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo controlled, randomized trial. Two arms, one is the intervention arm which will receive EMLA cream and local anesthesia infiltration while the control arm will receive local anesthesia infiltration and a control, lotion cream.
Who Masked: Participant, Care Provider
Masking Description: The surgeon and patient are both blinded to which cream is being utilized, whether it be EMLA, or a control cream. Investigators and study personelle are not blinded to this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm - EMLA cream (Experimental): This arm will receive EMLA cream 30 minutes prior to their procedure, applied to the scrotum. The patient is blinded to which cream they have received and this cream is removed prior to entering the procedural suite.
  Interventions: Drug: Eutectic mixture of local anesthetics (EMLA; Astra Pharmaceutical Products Inc., Westborough, MA)
- Control arm - Control cream (Placebo Comparator): This arm will receive lotion cream 30 minutes prior to their procedure, applied to the scrotum. The patient is blinded to which cream they have received and this cream is removed prior to entering the procedural suite.
  Interventions: Other: Control cream

INTERVENTIONS:
Drug: Eutectic mixture of local anesthetics (EMLA; Astra Pharmaceutical Products Inc., Westborough, MA) — The intervention is the utilization of EMLA cream, a topical anesthetic to determine if this reduces pain with local anesthesia infiltration, and for overall procedural pain
  Other Names: EMLA
  Arms: Intervention arm - EMLA cream
Other: Control cream — This intervention will be for the control group, a simple lotion cream.
  Other Names: Moisturizing cream
  Arms: Control arm - Control cream

SUMMARY:
Scrotal, urologic surgery has traditionally been conducted in the hospital setting, typically with the use of sedation, spinal anesthesia or general anesthesia. There has been a recent push to move certain scrotal urologic surgeries out of the hospital operating room into a ambulatory, outpatient basis with recent literature demonstrating this in many centers. The use of local anesthesia alone poses numerous benefits. The investigators wish to compare patients who are undergoing invasive scrotal surgery under local anesthetic to those who additionally have a topical anesthetic cream (EMLA) applied to the scrotum to determine if this further increases patient tolerability of these procedures.

DETAILED DESCRIPTION:
The current standard of care for patients undergoing the majority of urologic procedures is to administer general or spinal anesthesia. The use of general or spinal anesthesia can lead to several complications, long wait times, higher costs associated with the operating. While office-based surgical procedures under local anesthesia can have additional benefits aside from avoiding adverse effects of spinal or general anesthesia, such as ability to communicate, improved convenience, and absence of extended post-op recovery. In one particular study, patients who were surveyed were overwhelmingly satisfied with office-based procedures, and often perceived office-based procedures as less invasive and safer. Urologic care has much to gain from expanding the use of procedures performed under local anesthetic in an ambulatory setting to address the above problems.

Although local anesthetic can be quite effective, needle phobia and negative experiences associated with it can be a common experience. In addition to the fear associated with injection, the traditional local anesthetic injection can also be associated with pain and trauma to the infiltrated site. EMLA (Eutectic Mixture of Local Anesthetic) is a topic anesthetic cream that has in various office based urology procedures. Its use and potential benefits has been seen in a few studies for use in no-scalpel vasectomy, circumcision, metatomy, and more. However its use in more involved/invasive andrology and male-infertility procedures such as hydrocelectomy, penile plications, and others remain poorly studied thus far. Anecdotally, use of EMLA cream as an adjunct to our local anesthetic protocol demonstrated good efficacy in pain control and patient tolerability.

As such, the investigators wish to perform a prospective randomized controlled study at the Manitoba Men's Health Clinic to assess whether or not the use of EMLA cream and local anesthetic nerve block is associated with improved pain tolerance than local anesthetic alone. If our hypothesis provides true, further implementation of EMLA cream in office based andrology and male-infertility procedures may provide better pain control and overall experience for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing hydrocelectomy, spermatocelectomy, epididymectomy, testicular biopsy, scrotal lesion or cyst excision under local anesthesia alone were included.

Exclusion Criteria:

* Patients were excluded if their procedure was to be performed with sedatives (e.g., inhaled nitrous oxide gas, oral, or IV sedation) or did not provide consent to be randomized

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain with local anesthetic infiltration | Immediately post-infiltration, intraoperatively
  Using a visual analogue pain scale [range 0-10; 0 = no pain, 10 = maximal pain], pain will be assessed as reported by the patient when the local anesthetic injection is administered
Procedural pain | Immediately post-operation
  Using a visual analogue pain scale [range 0-10; 0 = no pain, 10 = maximal pain], pain will be assessed as reported by the patient post-operatively to determine their pain

CONTACTS AND LOCATIONS:
Locations (1):
- Men's Health Clinic Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Chung D, Bal DS, Morra M, Shah J, Fidel MG, Dhillon H, Van Heerden H, Nayak JG, Patel P. Efficacy of EMLA for Office-based Andrology Procedures Under Local Anesthesia: A Randomized Control Trial. Urology. 2024 Oct;192:6-11. doi: 10.1016/j.urology.2024.07.004. Epub 2024 Jul 5. PMID 38972394